CLINICAL TRIAL: NCT00168376
Title: A Randomised Double-Blind Trial of Targeted Repetitive Transcranial Magnetic Stimulation in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 57/04
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Last update posted 2007-04-16 (Estimated); Status verified 2007-04

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
The study will involve a 3-week (15 session) randomized double-blind clinical trial of two repetitive transcranial magnetic stimulation (rTMS) conditions in patients with treatment resistant depression. rTMS site selection will be localized from structural MRI scans.

The patients will be randomized to one of two conditions

1. rTMS targeted to the border of Brodmann area 46 and Brodmann area 9,
2. rTMS targeted to premotor cortex (this condition will act as the non-dorsolateral prefrontal cortex targeted control).

DETAILED DESCRIPTION:
The outcome measure used is the MADRS (Montgomery-Asberg Depression Rating Scale). This is administered at baseline and on a fortnightly basis. At study end response criteria is defined as a 50% reduction in total MADRS score and remission defined as a MADRS score of less than or equal to 10.

Other outcome measures administered fortnightly are: BPRS (Brief Psychiatric Rating Scale), CORE (measure of melancholic symptoms), BDI (Beck Depression Inventory), CGI (Clinical Global Impression Scale), GAF (Global Assessment of Functioning Scale). A cognitive battery is also administered.

Inclusion Criteria:

* Moderate to severe depressive symptoms as indicated as MADRS >20
* Failure to respond to a minimum of two antidepressant medications
* No increase or initiation of new antidepressant therapy in the four weeks prior to entering the trial Exclusion Criteria
* Have an unstable medical condition, neurological disorder or any history of seizure disorder or are currently pregnant or lactating
* Previous brain injury or surgery, any metal clips, plates or other metal items in the head, cardiac pacemaker
* In the opinion of the investigator, are a sufficient suicide risk to require immediate electroconvulsive therapy
* Have a current DSMIV diagnosis of substance abuse or dependence disorder, a diagnosis of a personality disorder or another axis 1 disorder

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe depressive symptoms as indicated as MADRS >20
* Failure to respond to a minimum of two antidepressant medications
* No increase or initiation of new antidepressant therapy in the four weeks prior to entering the trial

Exclusion Criteria:

* Have an unstable medical condition, neurological disorder or any history of seizure disorder or are currently pregnant or lactating
* Previous brain injury or surgery, any metal clips, plates or other metal items in the head, cardiac pacemaker
* In the opinion of the investigator, are a sufficient suicide risk to require immediate electroconvulsive therapy
* Have a current DSMIV diagnosis of substance abuse or dependence disorder, a diagnosis of a personality disorder or another axis 1 disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-07; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The outcome measure used is the MADRS (Montgomery-Asberg Depression Rating Scale). This is administered at baseline and on a fortnightly basis.

SECONDARY OUTCOMES:
Other outcome measures administered fortnightly are: BPRS (Brief Psychiatric Rating Scale), CORE (measure of melancholic symptoms), BDI (Beck Depression Inventory), CGI (Clinical Global Impression Scale), GAF (Global Assessment of Functioning Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Fitzgerald, MBBS, PhD, Principal Investigator — Alfred Psychiatry Research Centre
Locations (1):
- Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Fitzgerald PB, Hoy K, McQueen S, Maller JJ, Herring S, Segrave R, Bailey M, Been G, Kulkarni J, Daskalakis ZJ. A randomized trial of rTMS targeted with MRI based neuro-navigation in treatment-resistant depression. Neuropsychopharmacology. 2009 Apr;34(5):1255-62. doi: 10.1038/npp.2008.233. Epub 2009 Jan 14. PMID 19145228